CLINICAL TRIAL: NCT06267976
Title: Validation of the ProSomnus® RPMO2 Pulse Oximeter Device
Brief Title: Validation of the ProSomnus® RPMO2 Device
Status: Completed | Type: Observational
Sponsor: ProSomnus Sleep Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: REB23-1003
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: pulse oximeter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Healthy volunteers: Health adult volunteers will undergo a controlled desaturation to collect data for validation of the RPMO2 device.
  Interventions: Device: ProSomnus RPMO2

INTERVENTIONS:
Device: ProSomnus RPMO2 — The ProSomnus RPMO2 device is an intraoral reflectance pulse oximeter.

SUMMARY:
The purpose of the study is to:

1. Evaluate the SpO2 accuracy of the oximeter component of the ProSomnus RPMO2 Device during non-motion conditions over the range of 70-100% SaO2 by comparison to SaO2 values determined by arterial blood sample specimen analyzed by a CO-oximeter.
2. Evaluate the pulse rate performance simultaneously collected over the SpO2 range.

DETAILED DESCRIPTION:
Testing will be performed with participants semi-recumbent, under non-motion conditions. SpO2 accuracy of the test device will be determined by a controlled desaturation study with measurements taken over the full range of SaO2 values for which accuracy is to be claimed +3% of the lower value and -3% of the upper value. Participants will be desaturated to achieve six plateaus between 100-70% SaO2.

Arterial blood draws within the hypoxic plateaus will be performed, with draws occurring no less than 30 seconds after reaching a plateau and no less than 20 seconds apart. Five blood draws will be taken at each plateau. Plateaus will be determined using the reference transmittance pulse oximeter and are defined as a change in SpO2 on the reference pulse oximeter of no more than 1% over a duration of 20 seconds. Sampling will not continue if the blood oxygen saturation destabilizes between blood draws.

Time in low O2 saturation decades (i.e., 70-80% and 80-90%) will be limited to the minimum amount of time required to obtain test data and will not exceed 10 minutes. The saturation level at each plateau and the number of plateaus may vary among participants. Arterial pressure, ECG, heart rate, EtCO2, respiratory rate, and FiO2 will be monitored during testing. Extra samples may be collected at the discretion of the PI. The controlled desaturation protocol is expected to take approximately 30 to 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 18 and < 50 years.
* In good health with no evidence of medical problems.
* Ability to provide informed consent and willingness to comply with the study procedures.
* Ability to undergo controlled hypoxemia to the levels outlined in the desaturation profile.
* Adequate dentition for an oral appliance.
* Ability to breathe through the nose comfortably.

Exclusion Criteria:

* Obesity (BMI > 40 kg/m2).
* Known history of heart, lung, kidney, or liver disease.
* Diagnosis of asthma or sleep apnea.
* Diagnosis of diabetes.
* Presence of a clotting disorder.
* Presence of hemoglobinopathy or history of anemia that, in the opinion of the PI, makes the individual unsuitable for participation.
* Current smoker.
* History of fainting or vasovagal response.
* History of sensitivity to local anesthesia.
* Unacceptable collateral circulation based on exam (Allen's test).
* Pregnancy or lactation.
* Resting heart rate > 120 bpm.
* Systolic BP > 150, diastolic BP > 90.
* Carboxyhemoglobin level > 3%.
* Presence of any other condition that, in the opinion of the PI, makes the individual unsuitable for participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include volunteers who have previously been determined to be healthy enough for the study and who have signed an informed consent form and met the eligibility criteria.
  A minimum of 10 healthy participants will be recruited to complete the test protocol. A minimum of two participants or 15% of the participant pool (whichever is larger) will have Fitzpatrick Skin type IV, V, or VI (i.e., darkly pigmented skin).
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
SpO2 accuracy | 2 hours
  Root-mean-square (Rms) ± 3.5 [% SpO2] over the range of 70 to 100% SaO2
Pulse rate accuracy | 2 hours
  Rms within ± 3 [1/min] over the claimed range

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No